CLINICAL TRIAL: NCT03064204
Title: The Pathogenesis of OSA in People Living With HIV
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Center For AIDS Research Creative and Novel Ideas in HIV Research (CFAR CNIHR) (Unknown)
Responsible Party: Principal Investigator, Robert L. Owens, Associate Physician, University of California, San Diego
Other Study IDs: UCSD 161299
Record Dates: First submitted 2017-02-17; First posted 2017-02-24 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea; HIV/AIDS
MeSH Terms: conditions — Sleep Apnea, Obstructive; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSA+CPAP+HIV+: Individuals (40 years or older) diagnosed with OSA and using CPAP, also with HIV treated to viral suppression.
- OSA+CPAP+HIV-: Individuals (40 years or older) diagnosed with OSA and using CPAP.

SUMMARY:
The purpose of this study is to help us understand how HIV and/or Anti-Retroviral Therapy (ART) may predispose individuals to Obstructive Sleep Apnea (OSA). The traditional risk factors for OSA are weight and age. However, people living with HIV on ART seem to have OSA even when they are thin and young. The study involves a detailed physiological sleep study and an MRI of the head and neck to understand the underlying cause of OSA in those with and without HIV.

DETAILED DESCRIPTION:
Participants who have sleep apnea and are using positive airway pressure (PAP) with and without HIV will be enrolled if they otherwise meet all the inclusion criteria, and none of the exclusion criteria.

Subjects will undergo two overnight sleep studies (polysomnograms, PSGs) and a MRI scan of the upper airway. The first sleep study will evaluate the severity of sleep disordered breathing and will be identical to a clinical PSG. The second sleep study will measure the physiological traits most important for OSA, such as upper airway anatomy, control of breathing, sleep stability, and upper airway muscle activation. These measurements are performed while subjects sleep using PAP, but the PAP level is adjusted during the night, and the subject's response is measured. The MRI scan will be of the head and neck and will occur during the evening time. Subjects will be encouraged to sleep during this portion of the study, as well.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with physician-diagnosed OSA who have been prescribed CPAP Ages >= 40 years old
* BMI 20 - 35 kg/m2
* For HIV group: physician diagnosis of HIV and viral suppression

Exclusion Criteria:

* Not compliant with CPAP (by Medicare criteria, e.g. ≥4 hours per night on 70% of nights during a consecutive 30-day period via direct download or visual inspection of usage data).
* Use of medication that affects the traits, e.g. narcotics or sedative-hypnotics
* Any cardiovascular, pulmonary or renal disease other than well controlled hypertension or asthma.
* Pregnancy
* Currently smoking
* Any respiratory disorder other than OSA or well controlled asthma
* contraindication to MRI

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women with physician-diagnosed OSA who have been prescribed and are using positive airway pressure (e.g. CPAP). Also, men and women with physician-diagnosed HIV who achieved viral suppresion.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Upper airway collapsibility (Vpassive) | Night 2 (Visit 2 - to occur within 6 weeks of enrollment)
  Upper airway collapsibility, as assessed by rapid withdrawal of PAP

SECONDARY OUTCOMES:
Upper airway muscle responsiveness | Night 2 (Visit 2 - to occur within 6 weeks of enrollment)
  As assessed by rapid withdrawal of PAP
Pharyngeal fat pad thickness | MRI study (Visit 3 - to occur within 6 weeks of enrollment)
  As measured by MRI of the head and neck

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

REFERENCES:
- [Background] Darquenne C, Hicks CB, Malhotra A. The ongoing need for good physiological investigation: obstructive sleep apnea in HIV patients as a paradigm. J Appl Physiol (1985). 2015 Jan 15;118(2):244-6. doi: 10.1152/japplphysiol.00656.2014. Epub 2014 Aug 21. No abstract available. PMID 25150224
- [Background] Patil SP, Brown TT, Jacobson LP, Margolick JB, Laffan A, Johnson-Hill L, Godfrey R, Johnson J, Reynolds S, Schwartz AR, Smith PL. Sleep disordered breathing, fatigue, and sleepiness in HIV-infected and -uninfected men. PLoS One. 2014 Jul 3;9(7):e99258. doi: 10.1371/journal.pone.0099258. eCollection 2014. PMID 24991815